CLINICAL TRIAL: NCT02362217
Title: A Phase I Study to Evaluate the Safety and Immunogenicity of Simultaneous Prime-Boost Immunisations With Candidate HCV and HIV-1 Vaccines, AdCh3NSmut1 / ChAdV63.HIVconsv and MVA-NSmut / MVA.HIVconsv, in Healthy Volunteers
Brief Title: A Study to Assess the Safety of HIV and Hep C Vaccine Candidates When Given Separately or in Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: ReiThera Srl (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEACHI-04
Record Dates: First submitted 2014-11-06; First posted 2015-02-12 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Hepatitis C Infection; HIV Infection
MeSH Terms: conditions — Hepatitis C; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Interventions: AdCh3NSmut1, MVA-NSmut. Administration schedule: 1 dose AdCh3NSmut1 2.5 x 10^10 vp at week 0 and 1 dose MVA-NSmut 2 x 10^8 pfu at week 8.
  Subjects: 8 healthy volunteers.
  Interventions: Biological: AdCh3NSmut1; Biological: MVA-NSmut
- Group 2 (Experimental): Interventions: ChAdV63.HIVconsv, MVA.HIVconsv. Administration schedule: 1 dose ChAdV63.HIVconsv 5 x 10^10 vp at week 0 and 1 dose MVA.HIVconsv 2 x 10^8 pfu at week 8.
  Subjects: 8 healthy volunteers.
  Interventions: Biological: ChAdV63.HIVconsv; Biological: MVA.HIVconsv
- Group 3 (Experimental): Interventions: AdCh3NSmut1, MVA-NSmut, ChAdV63.HIVconsv, MVA.HIVconsv. Administration schedule: 1 dose AdCh3NSmut1 2.5 x 10^10 vp and 1 dose ChAdV63.HIVconsv 5 x 10^10 vp at week 0, and 1 dose MVA-NSmut 1 x 10^8 pfu and 1 dose MVA.HIVconsv 1 x 10^8 pfu at week 8.
  Subjects: 16 healthy volunteers.
  Interventions: Biological: AdCh3NSmut1; Biological: MVA-NSmut; Biological: ChAdV63.HIVconsv; Biological: MVA.HIVconsv

INTERVENTIONS:
Biological: AdCh3NSmut1 — Genetic vaccine against Hepatitis C virus infection
  Arms: Group 1; Group 3
Biological: MVA-NSmut — Genetic vaccine against Hepatitis C virus infection
  Arms: Group 1; Group 3
Biological: ChAdV63.HIVconsv — Genetic vaccine against HIV-1 infection
  Arms: Group 2; Group 3
Biological: MVA.HIVconsv — Genetic vaccine against HIV-1 infection
  Arms: Group 2; Group 3

SUMMARY:
This study is aimed at assessing the safety of candidate Hepatitis C vaccines AdCh3NSmut/MVA-NSmut and HIV vaccines ChAdV63.HIVconsv/MVA.HIVconsv when administered separately or in combination to healthy volunteers. The study also aims to assess the cellular immune response generated by these vaccines when administered as mentioned above.

DETAILED DESCRIPTION:
Hepatitis C and HIV are both widespread pathogens. By the end of 2010, there were 2.3 million people in Europe living with HIV, over half of whom were coinfected with the Hepatitis C virus (HCV). Although vaccination is the optimal method of preventing infection, it has proved extremely difficult to develop an effective vaccine against HIV and HCV due to the enormous variation in strains around the world. This is caused by the extraordinary ability of the viruses to change their genetic material.

Researchers at the University of Oxford have developed novel candidate vaccines against HIV ('HIV.consv') and HCV ('NSmut'). These vaccines have been inserted into the carrier viruses Chimpanzee Adenovirus (ChAd or AdCh) and modified vaccinia virus Ankara (MVA), both of which have excellent safety records. The aim of this study is to test for the first time the response of the immune system when vaccines to both HIV and HCV are given together.

During this study, 32 healthy adults aged 18 to 50 years will be recruited into one of three groups to receive either two or four intramuscular injections over a period of two months. All participants will be followed up for a further six months (12 visits in total).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, as assessed by medical history, physical examination and laboratory tests
* Aged at least 18 years on the day of screening and no greater than 50 years on the day of the first vaccination
* Resident in or easy access to the trial site for the duration of the study
* Available for follow-up for the planned duration of the study
* Able and willing (in the Chief Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females, willingness to practice continuous effective contraception from screening until 4 months after the last immunisation.
* All female volunteers must be willing to undergo urine pregnancy tests at the time points specified in the Schedule of Procedures and must have a negative pregnancy test on the day(s) of vaccination
* For sexually active men, willingness to use an approved method of contraception until four months after the last vaccination
* Agreement to refrain from blood donation during the course of the study
* In the opinion of the Chief Investigator or designee, the volunteer has understood the information provided. Written informed consent must be given before any study-related procedures are performed
* Willing to undergo HCV/HIV-1 testing, counselling and receive test results

Exclusion Criteria:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of a recombinant simian adenoviral vaccine
* Receipt of any investigational HIV-1 or HCV vaccine within the last 6 years
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Receipt of live attenuated vaccine within the previous 60 days or planned receipt within 60 days after vaccination with the IMP
* Receipt of other vaccine, including influenza vaccine, within the previous 14 days or planned receipt within 14 days after vaccination with the IMP
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressive medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* History of clinically significant contact dermatitis
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug use
* Reported high-risk behaviour for HIV-1 / HCV infection
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for HIV-1 (antibodies to HIV-1) at screening
* Seropositive for hepatitis C virus (antibodies to HCV) at screening
* Any other clinically significant acute or chronic medical condition that is considered unstable/progressive, or in the opinion of the Chief Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the protocol
* Vulnerable subjects (according to ICH GCP)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Safety of administering simultaneous HCV/HIV-1 prime-boost vaccinations, as measured by the proportion of volunteers who develop a grade 3 or 4 local or systemic reaction | Actively collected throughout the study until 6 months after the last vaccination
  Proportion of volunteers who develop a grade 3 or 4 local reaction Proportion of volunteers who develop a grade 3 or 4 systemic reaction

SECONDARY OUTCOMES:
Cellular immune response generated by simultaneous HCV/HIV-1 prime-boost vaccinations, as determined by analysing changes in the magnitude or quality of HCV and HIV-1-specific cellular immune responses. | Actively collected throughout the study until 6 months after the last vaccination
  Immunogenicity determined by analysing changes from baseline in the magnitude or quality of HCV and HIV-1-specific cellular immune responses. These will be detected using several standardised assays. The primary outcome measure for immunogenicity will be the development of T cell responses to HCV and HIV-1 epitopes, as determined by IFN-ɣ ELISpot assay. In addition, several exploratory immunology assays (including but not limited to intracellular cytokine staining, phenotype, viral suppression in vitro) will be developed and used.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Dorrell, Prof., Study Chair — University of Oxford; Ellie Barnes, Prof., Principal Investigator — University of Oxford; Tomas Hanke, Prof., Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hartnell F, Brown A, Capone S, Kopycinski J, Bliss C, Makvandi-Nejad S, Swadling L, Ghaffari E, Cicconi P, Del Sorbo M, Sbrocchi R, Esposito I, Vassilev V, Marriott P, Gardiner CM, Bannan C, Bergin C, Hoffmann M, Turner B, Nicosia A, Folgori A, Hanke T, Barnes E, Dorrell L. A Novel Vaccine Strategy Employing Serologically Different Chimpanzee Adenoviral Vectors for the Prevention of HIV-1 and HCV Coinfection. Front Immunol. 2019 Jan 18;9:3175. doi: 10.3389/fimmu.2018.03175. eCollection 2018. PMID 30713538